CLINICAL TRIAL: NCT00816283
Title: BMS CA180157: A Phase I Combination Study of Dasatinib Plus Vorinostat in Accelerated Phase, Chronic Phase Refractory to Second Line Therapy or Blast Crisis Chronic Myelogenous Leukemia (CML), and in Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Dasatinib and Vorinostat in Treating Patients With Accelerated Phase or Blastic Phase Chronic Myelogenous Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08047; P30CA033572 (NIH); CHNMC-08047; CDR0000631569 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; Philadelphia chromosome positive adult precursor acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; Vorinostat; Cytogenetic Analysis; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dasatinib — 50 mg orally 2 times per day or 140 mg orally one time per day
Drug: vorinostat — 100 mg orally 2 times per day
Genetic: cytogenetic analysis — Performed at the end of cycle two of treatment and every six cycles for patients with accelerated CML and every 3 cycles for patients with blast crisis or Ph+ ALL
Genetic: gene expression analysis — Bone marrow aspirate obtained pre-treatment, at first scheduled bone marrow assay and at relapse. Peripheral blood drawn pre-therapy, day +14 of first treatment cycle and at relapse.
Genetic: mutation analysis — Performed at baseline and at every bone marrow analysis on peripheral blood
Genetic: reverse transcriptase-polymerase chain reaction — Peripheral blood drawn prior to starting Vorinostat on Day 1 and on Day 14 of treatment
Other: flow cytometry — Performed at the end of cycle two of treatment and every six cycles for patients with accelerated CML and every 3 cycles for patients with blast crisis or Ph+ ALL
Other: laboratory biomarker analysis — Performed pre-treatment and day +14 of treatment

SUMMARY:
RATIONALE: Dasatinib and vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving dasatinib together with vorinostat may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of dasatinib when given together with vorinostat in treating patients with accelerated phase or blastic phase chronic myelogenous leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To define the maximum tolerated dose of dasatinib and vorinostat in patients with accelerated phase or blastic phase chronic myelogenous leukemia or Philadelphia chromosome-positive acute lymphoblastic leukemia.
* To assess the toxicity of this regimen in these patients.
* To assess, preliminarily, the efficacy of this regimen in these patients.

Secondary

* To perform correlative studies relevant to this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral dasatinib twice daily on days 1-21 and oral vorinostat twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspiration and blood sample collection periodically for correlative laboratory studies. Samples are assessed by RT-PCR for DNA damage response and proapoptotic elements (GADD45, FANC, and FOXO3A); cytogenetic analysis; flow cytometry; mutation analysis of bcr-abl; and gene expression array analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Chronic myelogenous leukemia meeting 1 of the following criteria:

    * In accelerated phase, defined by the presence of ≥ 1 of the following:

      * At least 15% but < 30% blasts in peripheral blood and/or bone marrow
      * At least 30% blasts plus promyelocytes in peripheral blood or bone marrow (providing that < 30% blasts are present in bone marrow)
      * At least 20% basophils in peripheral blood
      * Platelet count < 100,000/mm³ (unrelated to therapy) OR platelet count > 100,000/mm³ and unresponsive to therapy
      * Cytogenetic evidence of clonal evolution
      * Increasing spleen size and increasing WBC count and unresponsive to therapy
    * In blastic phase (blast crisis), defined by the presence of ≥ 1 of the following:

      * At least 30% blasts in peripheral blood and/or bone marrow
      * Extramedullary infiltrates of leukemic cells (other than liver or spleen involvement)
  * Philadelphia chromosome-positive acute lymphoblastic leukemia meeting any of the following criteria:

    * Newly diagnosed or relapsed disease
    * Previously treated with chemotherapy, stem cell transplantation, or tyrosine kinase inhibitors (TKIs)
* No active CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin < 2.0 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Serum sodium, potassium, magnesium, phosphate, and calcium ≥ lower limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 4 weeks after discontinuation of study drug
* Able to take oral medication
* No active post-transplantation-related infections (e.g., fungal or viral infection)
* No active acute graft-versus-host disease (GVHD) of any grade
* No chronic GVHD (other than mild skin, oral, or ocular GVHD not requiring systemic immunosuppression)
* No other malignancy that required radiotherapy or systemic treatment within the past 5 years
* No concurrent medical condition that may increase the risk of toxicity, including pleural or pericardial effusion of any grade
* No cardiac conditions, including any of the following:

  * Uncontrolled angina, congestive heart failure, or myocardial infarction within the past 6 months
  * Diagnosed congenital long QT syndrome
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Prolonged QTc interval (i.e., QTc > 450 msec) on baseline EKG
* No hypokalemia or hypomagnesemia that cannot be corrected prior to dasatinib administration
* No history of significant bleeding disorder unrelated to cancer, including any of the following:

  * Diagnosed congenital bleeding disorder (e.g., von Willebrand's disease)
  * Acquired bleeding disorder diagnosed within the past year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (i.e., within the past 3 months) significant gastrointestinal bleeding
* No prisoners or individuals who are compulsorily detained (i.e., involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior HDAC inhibitors or compounds with HDAC inhibitor-like activity (e.g., valproic acid) as anti-tumor therapy

  * Prior valproic acid for the treatment of seizures allowed provided it was not given within the past 30 days
* Prior allogeneic stem cell transplantation allowed
* More than 4 weeks since prior chemotherapy other than TKI (6 weeks for nitrosoureas and mitomycin)
* More than 2 weeks since prior radiotherapy
* At least 7 days since prior and no concurrent Category I drugs that are generally accepted to have a risk of causing Torsades de pointes, including any of the following:

  * Quinidine, procainamide, or disopyramide
  * Amiodarone, sotalol, ibutilide, or dofetilide
  * Erythromycin or clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, or pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, or lidoflazine
* At least 7 days since prior and no concurrent medications that directly and durably inhibit platelet function, including any of the following:

  * Aspirin or aspirin-containing combinations, clopidogrel, or dipyridamole
  * Tirofiban, epoprostenol, eptifibatide, cilostazol, abciximab, ticlopidine, or cilostazol
* At least 5 days since prior and no concurrent St. John's wort
* No IV bisphosphonates during the first 8 weeks of dasatinib therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 21 days after the beginning of treatment
Toxicity as assessed by NCI CTCAE v3.0 | 21 days from the beginning of the last course of treatment
Response rate | One year after treatment completion
Objective tumor response | One year after treatment completion
Survival | One year after treatment completion
Time to treatment failure | One year after treatment completion
Duration of response | One year after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: David Snyder, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California